CLINICAL TRIAL: NCT07110636
Title: A Prospective Randomized Basket Trial Evaluating the Clinical Utility of Plasma-based Microbial Cell-free Metagenomic Sequencing for Diagnosis and Management of Suspected Infections in Adult Immunocompromised Outpatients
Brief Title: Microbial Cell-free Metagenomic Sequencing for Suspected Infections in Adult Immunocompromised Outpatients
Acronym: OPTIMUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karius, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KAR-0025
Record Dates: First submitted 2025-06-17; First posted 2025-08-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Infection; Infections, Bacterial; Infections, Fungal; Infection Viral; Parasitic Disease
Keywords: Karius; Karius Spectrum; Infection detection; metagenomic testing; Pathogen detection; Bacterial Infection; Fungal Infection; Parasitic Infection; Viral Infection
MeSH Terms: conditions — Infections; Bacterial Infections; Mycoses; Virus Diseases; Parasitic Diseases

STUDY DESIGN:
Intervention Model Description: Both the interventional group and control group will undergo a blood draw. The interventional group will receive Karius Spectrum test results. The control group will not receive Karius Spectrum test results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): This arm will receive Karius Spectrum test results.
  Interventions: Diagnostic Test: Metagenomic plasma-based test for agnostic pathogen detection
- Control (No Intervention): This arm will not receive Karius Spectrum test results.

INTERVENTIONS:
Diagnostic Test: Metagenomic plasma-based test for agnostic pathogen detection — Karius Spectrum metagenomic plasma-based test.
  Arms: Interventional

SUMMARY:
This clinical trial is designed to evaluate if adding the Karius Spectrum™ plasma test to usual care diagnostic tests, compared to usual care testing alone, among immunocompromised participants presenting with suspected infection in the outpatient setting leads to faster infection diagnosis and treatment. Participants will give a blood sample one time to be used for the testing. Information about the participant's illness and any treatments within 30 days following enrollment will be recorded.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled interventional trial designed to evaluate the clinical utility and effectiveness of adding the Karius Spectrum™ plasma test to usual care diagnostic tests, compared to usual care testing alone, among immunocompromised participants presenting with suspected infection in the outpatient setting.

The study is structured as a basket trial to enable the efficient evaluation of Karius Spectrum across multiple high-risk clinical populations with shared unmet diagnostic and management needs. The basket protocol outlines core trial elements applicable to all cohorts-including high-level objectives, study design, statistical framework, and operational procedures-while cohort-specific sub-protocols provide detailed rationale, objectives and endpoints, eligibility criteria, and contextual considerations tailored to each cohort. This design supports both pooled analyses across cohorts and subgroup assessments within distinct immunocompromised cohorts.

There are 2 cohorts: Cohort A, which is composed of patients that have had a solid organ transplant; and Cohort B, which is composed of patients that have a hematological malignancy, have had a stem cell transplant, or have undergone CAR-T therapy.

Karius Spectrum is a plasma-based microbial cell-free DNA (mcfDNA) metagenomic sequencing test for agnostic detection, identification, and quantification of more than 1,000 human microbial pathogens (i.e., microorganisms), including bacteria, DNA-based viruses, fungi, and parasites, potentially causing disease anywhere in the body. This test is intended for use in the diagnosis and management of suspected infections.

ELIGIBILITY:
Inclusion Criteria:

* Basket Protocol* All participants must meet inclusion

  1. Age ≥18
  2. Included in one of the following immunocompromised groups: Solid organ transplant recipient (SOT) on chronic immunosuppression; Diagnosed with hematologic malignancy (HM) and/or recipient of a hematopoietic cell transplant (HCT); Diagnosed with a solid tumor and on specific types of active treatment; Recipient of drugs or novel biologics causing chronic immunosuppression; Diagnosed with an HIV infection; Diagnosed with inborn errors of immunity
  3. Treating provider suspects infection and plans to obtain usual care diagnostic testing for the suspected infection (i.e., microbiologic testing)
  4. Willing to provide research samples via blood draw
  5. Willing and able to provide informed consent
  6. Presenting for evaluation in the outpatient setting (includes telehealth)

     *For Participants enrolled in Sub-Protocol A- Solid Organ Transplant*

     All Sub-Protocol A subjects must meet the following:

  <!-- -->

  1. Solid organ transplant recipient on transplant immunosuppression Non-lung recipients must meet one or more of the following characteristics: <1 year from transplant; Augmented immunosuppression for suspected or confirmed rejection within the last 6 months; Confirmed systemic infection in last 6 months
  2. Suspected infection defined by one or more of the syndromes: Cardiac; Lower Respiratory; Gastrointestinal / Hepatobiliary; Genitourinary; Neurologic / Ophthalmologic; Skin / Soft tissue / musculoskeletal; Not Otherwise Specified
* For Participants enrolled in Sub-Protocol B- Hematological Malignancies and Transplant* All Sub-Protocol B subjects must meet the following:

  1. Is included in at least one of the following groups: Hematologic malignancy (leukemia, myelodysplastic syndrome, lymphoma, multiple myeloma) and at least one of the following: Received chemotherapy or other systemic anti-cancer therapy associated with immunosuppressive effects within 90 days (e.g., monoclonal antibodies associated with B-cell or plasma cell depletion, bi-specific t-cell engagers, BTK inhibitors, BCL-2 inhibitors, PI3K inhibitors) within the last 90 days Note: Checkpoint inhibitors are not included unless given in combination with an immunosuppressive agent; Relapsed disease with chemotherapy anticipated in 60 days; ANC <500 within the last 72 hours; Hypogammaglobulinemia IgG <400 within the last 30 days; Allogeneic stem cell transplant for any clinical indication and at least one of the following: Within 1-year post-transplant; On systemic immunosuppressive therapy for GVHD treatment or prophylaxis; Autologous stem cell transplant for hematologic malignancy and at least one of the following: Within 6 months post-transplant; ANC <500 within the last 72 hours; B cell and plasma cell targeted CAR-T therapy for hematologic malignancy and at least one of the following: Within 6 months of CAR-T cell infusion; CD4 T-cell <200 within the last 30 days; IgG < 400 within the last 30 days; ANC <500 within the last 72 hours; On systemic immunosuppressive therapy for CRS/ICANS
  2. Suspected infection defined by one or more of the syndromes: Cardiac; Lower Respiratory; Gastrointestinal / Hepatobiliary; Genitourinary; Neurologic / Ophthalmologic; Skin / Soft tissue / musculoskeletal; Not Otherwise Specified

Exclusion Criteria:

* Basket Protocol* All participants must not meet the following:

  1. Active symptoms are likely attributed to non-infectious causes.
  2. Any other clinically significant medical condition that, in the opinion of the treating provider, makes participation undesirable, including but not limited to severe psychiatric illness, etc.

     *For Participants enrolled in Sub-Protocol A- Solid Organ Transplant*

     All Sub-Protocol A subjects must not meet the following:

  <!-- -->

  1. Patients who have been previously evaluated (including via telehealth) for the same clinical signs and symptoms at this institution and pathogen-directed usual care (UC), diagnostic testing was ordered during that prior encounter, with one or more diagnostic test results still pending.
  2. Patients with a suspected or confirmed primary upper respiratory infection (e.g., viral pharyngitis, sinusitis, or uncomplicated bronchitis) unless there is clinical suspicion of a concurrent lower respiratory or systemic infection requiring further diagnostic evaluation.
* For Participants enrolled in Sub-Protocol B- Hematological Malignancies and Transplant* All Sub-Protocol B subjects must not meet the following:

  1. Patients that have been previously evaluated (including via telehealth) for the same clinical signs and symptoms at this institution and pathogen-directed usual care (UC) diagnostic testing was ordered during that prior encounter with one or more diagnostic tests results still pending.
  2. Patients with a suspected or confirmed primary upper respiratory infection (e.g., viral pharyngitis, sinusitis, or uncomplicated bronchitis) unless there is clinical suspicion of a concurrent lower respiratory or systemic infection requiring further diagnostic evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to Identification of a Pathogen Specific Etiology | The study sample will be collected within 24 hours of enrollment; participant information including usual care laboratory testing and treatments will be collected for 30 days following enrollment.
  For each cohort, to evaluate whether the addition of Karius Spectrum testing to usual care testing reduces the time to identification of a pathogen-specific etiology, compared to usual care testing alone, in participants with suspected infection in the outpatient setting.
Time to Pathogen-Directed Treatment | The study sample will be collected within 24 hours of enrollment; participant information including usual care laboratory testing and treatments will be collected for 30 days following enrollment.
  For each cohort, to evaluate whether the addition of the Karius Spectrum test to usual care testing reduces the time to pathogen-directed treatment compared to usual care testing alone.

SECONDARY OUTCOMES:
Duration of Antimicrobial Therapy | 30 days following enrollment.
  For each cohort, to evaluate whether the addition of Karius Spectrum testing to usual care reduces the total duration of antimicrobial therapy during the 30-day follow-up period, using data abstracted from the electronic medical record (e.g., medication administration records and provider documentation).
Percentage of participants receiving pathogen-directed treatment | 30 days following enrollment.
  For each cohort, to evaluate whether the addition of Karius Spectrum testing to usual care testing increases the proportion of participants ultimately receiving pathogen-directed treatment compared to usual care testing alone at specific time points (e.g., Day 3, Day 7, Day 14).
Time to Clinically Meaningful Detection (CMD) | The study sample will be collected within 24 hours of enrollment; participant information including usual care laboratory testing and treatments will be collected for 30 days following enrollment.
  For each cohort, to evaluate whether the addition of Karius Spectrum testing to usual care testing is associated with a reduction in time to clinically meaningful detection (CMD) compared to usual care testing alone. A CMD event is defined as the earliest identification of either (1) an etiological pathogen, or (2) a non-etiological pathogen that prompts a clinically meaningful action (e.g., treatment initiation, specialist referral, diagnostic escalation, or vascular access removal). Only the first qualifying CMD event per participant will be used for analysis.
Number of Adverse Events | All AEs/SAEs will be collected from the time of blood draw through Day 30.
  For all cohorts, the number of participants experiencing adverse events (AEs) and serious adverse events (SAEs) that are unexpected or related to the Karius Spectrum test or study procedures will be assessed. Events will be summarized by type, severity, and relationship to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kat Kwiatkowski, PhD, Principal Investigator — Karius, Inc.
Locations (6):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - Ochsner Medical Center, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Montefiore Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No